CLINICAL TRIAL: NCT03339661
Title: Secondary Prophylaxis After CMV Disease in Kidney Transplant Patients Targeted by γδ T
Brief Title: Secondary Prophylaxis After CMV Disease in Kidney Transplant Patients Targeted by γδ T Cells Immunomonitoring.
Acronym: SPARCKLING
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2016/40
Record Dates: First submitted 2017-11-03; First posted 2017-11-13 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Kidney Transplant Infection
Keywords: CMV infection; kidney transplant; γδ T cells monitoring
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1_ No proph treatment (Experimental): Patients will receive a curative treatment (ganciclovir or valganciclovir, drug administrated will depend on medical opinion) during 2 to 8 weeks. When CMV QNAT becomes regative, if γδ T cell expansion occurs, no secondary prophylaxis treatment will be introduce, and curative treatment stops.
  Interventions: Drug: Group 1_No proph treatment
- Group 2A_Proph treatment and γδ T cells expansion (Experimental): Patients will receive a curative treatment (ganciclovir or valganciclovir, drug administrated depends on medical opinion) during 2 to 8 weeks. When CMV QNAT becomes regative, if no γδ T cell expansion will occur, a secondary prophylaxis will be initiated during 3 months maximum. The occurrence of γδ T cells expansion during or at the end of secondary prophylaxis will define the group 2A.
  Interventions: Drug: Group 2A_Proph treatment and γδ T cell expansion
- Group 2B_Proph treatment and no γδ T cells expansion (Experimental): Patients will receive a curative treatment (ganciclovir or valganciclovir, drug administrated depends on medical opinion) during 2 to 8 weeks. When CMV QNAT becomes regative, if no γδ T cell expansion will occur, a secondary prophylaxis will be initiated during 3 months maximum. Patients who still not had γδ T cells expansion during or at the end of secondary prophylaxis will compose the group 2B.
  Interventions: Drug: Group 2B_Proph treatment and no γδ T cell expansion

INTERVENTIONS:
Drug: Group 1_No proph treatment — After the curative treatment of CMV infection until a negative CMV ADNemia, secondary prophylaxis with valganciclovir will be established based on the results of γδ T cells immunomonitoring. In this group, expansion of γδ T cell at the end curative treatment was detected, so secondary prophylaxis will not be started.
  Arms: Group 1_ No proph treatment
Drug: Group 2A_Proph treatment and γδ T cell expansion — After the curative treatment of CMV infection until a negative CMV ADNemia, secondary prophylaxis with valganciclovir will be established based on the results of γδ T cells immunomonitoring. In this group, γδ T cell expansion will not be detected, so secondary prophylaxis will be initiated in continue during 3 months maximum. The occurrence of γδ T cells expansion during or at the end of secondary prophylaxis will define the group 2A.
  Arms: Group 2A_Proph treatment and γδ T cells expansion
Drug: Group 2B_Proph treatment and no γδ T cell expansion — After the curative treatment of CMV infection until a negative CMV ADNemia, secondary prophylaxis with valganciclovir will be established based on the results of γδ T cells immunomonitoring. In this group, γδ T cell expansion will not be detected, so secondary prophylaxis will be initiated in continue during 3 months maximum. Patients who still not had γδ T cells expansion during or at the end of secondary prophylaxis will compose the group 2B.
  Arms: Group 2B_Proph treatment and no γδ T cells expansion

SUMMARY:
In kidney transplant patients, CMV infection remains the leading infectious cause of morbidity and mortality. Clinical and virological relapses are common and are involved in chronic graft dysfunction. To date, it is not certain that secondary prophylaxis allows reducing these relapses, although this prophylaxis is part of the current recommendations. Our team has recently shown that the expansion of γδ T cells in peripheral blood during CMV infection was correlated with the absence of virological and clinical relapses. Indeed, the absence of relapse was associated in 94.7% of cases with the presence of γδ T cells expansion while relapses occurred in about 90% of cases in the absence of γδ T cells expansion. These results suggest that the indication and duration of secondary prophylaxis after the curative treatment of CMV infection in kidney transplantation could be guided by the immune surveillance of γδ T cells.

DETAILED DESCRIPTION:
The study aim to demonstrate that the expansion of γδ T cells at the end of curative treatment predicts the absence of virological and clinical relapses. This is a pilot study that will be conducted in the transplant center of Bordeaux and Lyon. After the curative treatment of CMV infection until a negative CMV ADNemia, secondary prophylaxis with valganciclovir will be established based on the results of γδ T cells immunomonitoring:

(I) Secondary prophylaxis will not be started in patients with γδ T cell expansion at the end of curative treatment (group 1) (II) Secondary prophylaxis will be initiated in patients who have not γδ T cell expansion and will continue for 3 months maximum. The occurrence of γδ T cells expansion during or at the end of secondary prophylaxis will define the group 2A. Patients who still not had γδ T cells expansion during or at the end of secondary prophylaxis will compose the group 2B.

The primary outcome of this study will be to evaluate the occurrence of virological relapse, assessed by monitoring CMV ADNemia, at one year of a first CMV disease, in kidney transplant patients, with secondary prophylaxis based on the monitoring of γδ T cells.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old without weight or ethnicity criteria, kidney transplant.
* Patient affiliated or beneficiary of a social security scheme.
* Patient with symptomatic or non-symptomatic CMV infection requiring curative treatment with ganciclovir or valganciclovir.
* Free, informed and written consent signed by the participant and the investigator (at the latest, on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Resistance documented to antivirals.
* Hemodialysis patient.
* Number of polymorphonuclear neutrophils less than 500 / μL and / or number of platelets less than 25,000 / μL, and / or lower hemoglobin 8 g / dL.
* Contraindication to valganciclovir, including known hypersensitivity to valganciclovir and / or aciclovir and / or valaciclovir or ganciclovir or their excipients, known severe intolerance to valganciclovir or ganciclovir.
* Women of childbearing age without a negative pregnancy test at baseline and without effective contraception (estrogen-progestin, intrauterine device) throughout the study period and two months after cessation of the follow-up period.
* Nursing women.
* Men without mechanical contraception during treatment and for at least 90 days after treatment.
* Ongoing participation in another clinical trial evaluating a drug. Participation in an observational study will not be considered a contraindication.
* The patient's foreseeable inability to comply with planned visits in the protocol.
* Non-negativation of CMV PCR at 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Assessment of virological relapse occurence | 12 months after inclusion visit
  The primary outcome of this study will be to evaluate the occurrence of virological relapse, assessed by monitoring CMV ADNemia.

SECONDARY OUTCOMES:
Cumulative incidence of clinical recurrence | 12 months after inclusion visit
  Cumulative incidence of clinical recurrence defined by a positive CMV PCR associated with clinical and biological signs of CMV disease. This incidence is expressed as a percentage of the total number of patients with CMV infection included.
γδ T cells expansion dynamic | 12 months after the inclusion visit
  Description of the dynamics of γδ T cells expansion in all patients. At each visit, an immunophenotyping with analysis of the percentage of γδ T cells will be performed.
Cumulative incidence of clinical recurrence at discontinuation of prophylaxis. | 12 months after the inclusion visit
  These incidences will be expressed as a percentage of the total number of patients who have had CMV infection included. Recidivism will be collected by the investigating physician when observed during a follow-up visit.
Cumulative incidence of virological recurrence at discontinuation of prophylaxis. | 12 months after inclusion visit
  These incidences will be expressed as a percentage of the total number of patients who have had CMV infection included. Recidivism will be collected by the investigating physician when observed during a follow-up visit.
secondary prophylaxis duration | 12 months after inclusion visit
  The duration of the secondary prophylaxis is defined by the duration of treatment since the stop of the curative treatment until the stop of the prophylactic treatment.
Prophylaxis treatment savings evaluation | 12 months after inclusion visit
  Evaluation of prophylaxis treatment savings (compared to a one-month prophylaxis) by number of subject and average total duration (with standard deviation) of treatment.
Proportion of antiviral resistant infections | 12 months after inclusion visit
  the proportion of antiviral resistant infections confirmed by genotypic analysis (mutations UL97 and UL54) sought during recurrence in case of clinical suspicion.
GFR average | 12 months after inclusion visit
  GFR average and its standard deviation are estimated according to MDRD formula
Compliance rate | 12 months after inclusion visit
  The compliance rate will, be performed by a patient notebook.

CONTACTS AND LOCATIONS:
Overall Officials: Edouard LHOMME, Dr, Study Chair — USMR
Locations (2):
- France (2):
  - Hôpital Pellegrin - CHU de Bordeaux, Bordeaux
  - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon